CLINICAL TRIAL: NCT03436394
Title: Phase I, Open-label, Single Dose Study to Investigate the Effect of Renal Impairment on the Pharmacokinetics (PK) of Evobrutinib (M2951) Compared to Normal Renal Function in Male and Female Subjects
Brief Title: Effect of Renal Impairment on Evobrutinib Pharmacokinetics (PK)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Merck KGaA, Darmstadt, Germany (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: MS200527_0026; 2017-004102-18 (EudraCT Number)
Record Dates: First submitted 2018-02-06; First posted 2018-02-19 (Actual); Last update posted 2019-05-16 (Actual); Status verified 2019-05

CONDITIONS: Renal Impairment
Keywords: Renal Impairment; Evobrutinib; Pharmacokinetics
MeSH Terms: conditions — Renal Insufficiency | interventions — evobrutinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Evobrutinib: Normal Renal Function (Experimental): Subjects with estimated glomerular filtration rate (eGFR) greater than or equal to (>=) 90 milliliter per minute per 1.73 meter square (mL/min/1.73 m^2) will receive a single oral dose of evobrutinib under fasting conditions.
  Interventions: Drug: Evobrutinib
- Evobrutinib: Severe Renal Impairment (Experimental): Subjects with eGFR less than (<) 30 mL/min/1.73 m^2 will receive a single oral dose of evobrutinib under fasting conditions.
  Interventions: Drug: Evobrutinib
- Evobrutinib: Moderate Renal Impairment (Experimental): Subjects with eGFR >= to 30 mL/min/1.73 m^2 and < 60 mL/min/1.73 m^2 will receive a single oral dose of evobrutinib under fasting conditions.
  Interventions: Drug: Evobrutinib
- Evobrutinib: Mild Renal Impairment (Experimental): Subjects with eGFR >= to 60 mL/min/1.73 m^2 and < 90 mL/min/1.73 m^2 will receive a single oral dose of evobrutinib under fasting conditions.
  Interventions: Drug: Evobrutinib

INTERVENTIONS:
Drug: Evobrutinib — Subjects will be administered a single oral dose of evobrutinib under fasting conditions.
  Other Names: MSC2364447C; M2951

SUMMARY:
The study will investigate the PK and safety of evobrutinib in subjects with different degree of renal impairment as compared to subjects with normal renal function.

ELIGIBILITY:
Inclusion Criteria:

* Male and Female subjects with total body weight between 50.0 and 100.0 kilograms(kg) (inclusive) and body mass index (BMI) between 19.0 and 36.0 kg per meter square (inclusive) at the time of the screening examination
* For subjects with impaired renal function: Subjects must have an eGFR according to the Modification of diet in renal disease (MDRD) equation of less than 90 mL per minute at screening and the possibility of stratification to one of the groups and a stable renal function as defined by either: if the time interval between screening and dosing is greater than 10 days, two eGFR with the second estimate within 20% of prior value or historical records of stable function over the past 3 months if within 20 percentage of screening value and within 10 days of dosing
* Other protocol defined inclusion criteria could apply

Exclusion Criteria:

* History or presence of respiratory, gastrointestinal (including bariatric or other gastric surgeries, or other conditions that may affect drug absorption) hepatic (including hepatorenal syndrome), hematological, lymphatic, neurological (including seizures), cardiovascular (including ventricular dysfunction and congestive heart failure), psychiatric, musculoskeletal, genitourinary, immunological, dermatological, connective tissue diseases or disorders that may affect the safety of the subject.
* Clinical history of any autoimmune disorder
* Prior history of cholecystectomy or splenectomy, and any clinically relevant surgery within 6 months prior to Screening, which might interfere with the objectives of the study or the study procedures
* History of any malignancy except superficial basal cell carcinoma treated for curative intent may be allowed
* Other protocol defined exclusion criteria could apply

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2018-03-21 (Actual); Primary Completion 2019-02-22 (Actual); Study Completion 2019-02-22 (Actual)

PRIMARY OUTCOMES:
Area Under the Plasma Concentration-Time Curve From Time Zero to the Last Quantifiable Concentration (AUC 0-t) of Evobrutinib | Pre-dose up to 30 hours post-dose
Area Under the Plasma Concentration-Time Curve From Time Zero Extrapolated to Infinity (AUC 0-inf) of Evobrutinib | Pre-dose up to 30 hours post-dose
Maximum Observed Plasma Concentration (Cmax) of Evobrutinib | Pre-dose up to 30 hours post-dose

SECONDARY OUTCOMES:
Occurrences of Treatment-emergent Adverse Events (TEAEs) | Day 1 up to Day 6
Number of Subjects With TEAEs According to Severity | Day 1 up to Day 6
Number of Subjects With Clinically Significant Abnormalities in Vital Signs, Laboratory Parameters and 12-lead Electrocardiogram (ECG) Findings | Day 1 up to Day 6
  Number of subjects with clinically significant abnormalities will be reported.
Time to Reach the Maximum Plasma Concentration (tmax) of Evobrutinib | Pre-dose up to 30 hours post-dose
Time Prior to the First Measurable (Non-Zero) Concentration (t lag) of Evobrutinib | Pre-dose up to 30 hours post-dose
Terminal Rate Constant (λz) of Evobrutinib | Pre-dose up to 30 hours post-dose
Terminal Half-Life (t1/2) of Evobrutinib | Pre-dose up to 30 hours post-dose
Area Under the Plasma Concentration-Time Curve From Time Zero to 24 Hours After Dosing (AUC 0-24h) of Evobrutinib | Pre-dose up to 24 hours post-dose
Area Under the Plasma Concentration-Time Curve From Time Zero to 8 Hours After Dosing (AUC 0-8h) of Evobrutinib | Pre-dose up to 8 hours post-dose
Apparent Clearance (CL/f) of Evobrutinib | Pre-dose up to 30 hours post-dose
Apparent Volume of Distribution During Terminal Phase (Vz/f) of Evobrutinib | Pre-dose up to 30 hours post-dose
Amount of Unchanged Drug (Evobrutinib) Excreted in Urine During Collection Interval (0-8 hours) (Ae0-8h) | Pre-dose up to 8 hours post-dose
Fraction of Administered Drug (Evobrutinib) Excreted in Urine (fe) | Pre-dose up to 30 hours post-dose
Fraction of Unbound Drug (Evobrutinib) in the Plasma (fu) | Pre-dose up to 30 hours post-dose
Renal Clearance of Evobrutinib (CLR) | Pre-dose up to 30 hours post-dose
Non-Renal Clearance of Evobrutinib (CLNonR/f) | Pre-dose up to 30 hours post-dose

CONTACTS AND LOCATIONS:
Overall Officials: Medical Responsible, Study Director — Merck KGaA, Darmstadt, Germany
Locations (1):
- Please Contact the Merck KGaA Communication Center, Darmstadt, Germany